CLINICAL TRIAL: NCT06955325
Title: A Randomized, Phase III Umbrella Trial of Adjuvant Therapy Versus Observation in Completely Resected High-Risk Stage IA-IB Non-Small Cell Lung Cancer Based on Oncogenic Driver Mutations
Brief Title: Umbrella Trial of Adjuvant Therapy in Completely Resected High-risk Stage IA-IB NSCLC: Focus on Driver Mutations
Acronym: UPLIFT
Status: Not yet recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: The First Affiliated Hospital of Guangzhou Medical University (Other)
Responsible Party: Principal Investigator, Jianxing He, Director, Head of Thoracic Surgery, Principal Investigator, Clinical Professor, The First Affiliated Hospital of Guangzhou Medical University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: UPLIFT
Record Dates: First submitted 2025-04-16; First posted 2025-05-02 (Actual); Last update posted 2025-05-06 (Actual); Status verified 2025-05

CONDITIONS: Non-Small Cell Lung Cancer
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung | interventions — icotinib; rezivertinib; ensartinib

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Adjuvant therapy (Experimental)
  Interventions: Drug: Icotinib; Drug: Rezivertinib; Drug: Ensartinib; Drug: Benmelstobart
- Observation (No Intervention)

INTERVENTIONS:
Drug: Icotinib — Oral icotinib tablets (125 mg) administered three times daily (TID) for up to 1 year or until disease recurrence or unacceptable toxicity. Icotinib is an EGFR tyrosine kinase inhibitor targeting EGFR-sensitizing mutations.
  Arms: Adjuvant therapy
Drug: Rezivertinib — Oral rezivertinib capsules (100 mg) taken once daily (QD) for up to 1 year or until disease recurrence or unacceptable toxicity. Rezivertinib is an EGFR tyrosine kinase inhibitor targeting EGFR-sensitizing mutations.
  Arms: Adjuvant therapy
Drug: Ensartinib — Oral ensartinib capsules (225 mg) taken once daily (QD) for up to 1 year or until disease recurrence or unacceptable toxicity. Ensartinib is an ALK/ROS1 tyrosine kinase inhibitor designed to inhibit ALK/ROS1 fusion-driven NSCLC.
  Arms: Adjuvant therapy
Drug: Benmelstobart — Intravenous infusion of bemosumab 1200 mg every 3 weeks (Q3W). Treatment continues for up to 4 cycles initially, and may be extended (maintenance) for up to 3 years or until disease recurrence or unacceptable toxicity. Bemosumab is a monoclonal antibody under investigation for immunotherapy in NSCLC.
  Arms: Adjuvant therapy

SUMMARY:
This study explores how adjuvant therapy affects survival in completely resected high-risk stage IA-IB NSCLC patients with different driver gene mutations.

DETAILED DESCRIPTION:
This study aims to evaluate whether tailored, targeted therapy or immunotherapy can effectively prevent cancer recurrence in patients with early-stage (stage IA-IB) non-small cell lung cancer (NSCLC) who have undergone complete surgical resection but are at high risk of recurrence. Based on each patient's specific driver gene mutation status (e.g., EGFR or ALK/ROS1) or wild-type status, participants will receive either targeted therapy or immunotherapy compared to routine follow-up (observation). The goal is to see if these approaches can improve disease-free survival and potentially reduce the risk of lung cancer recurrence.

ELIGIBILITY:
Inclusion Criteria:

* Age 18-75 years and able to provide written informed consent.
* Primary non-squamous NSCLC confirmed by pathology, with no brain metastases.
* Complete R0 surgical resection (lobectomy, segmentectomy, or pneumonectomy) of stage IA or IB NSCLC (AJCC 8th edition).
* High-risk disease (one or more): low differentiation, solid/micropapillary/complex glandular patterns, vascular invasion, visceral pleural invasion, alveolar space spread, or intermediate/high risk on 14-gene test.
* Documented driver gene status (EGFR mutation, ALK/ROS1 fusion, or wild-type) via postoperative tumor sample.
* ECOG performance status 0 or 1, with stable condition over the last two weeks.
* Surgery within 4-10 weeks before starting treatment, with full recovery.
* Adequate organ function as per protocol-defined labs.
* Negative pregnancy test (if applicable) and use of effective contraception during and 3 months after treatment.

Exclusion Criteria:

* Evidence of unresectable/metastatic NSCLC, incomplete resection (R1/R2), or wedge resection only.
* Prior systemic therapy (e.g., chemotherapy, targeted therapy, immunotherapy) for the current NSCLC.
* Major surgery (excluding lung cancer surgery) within 3 weeks before first study dose.
* Planned concurrent anti-cancer therapy (chemo, radiotherapy, or targeted therapy) during the study.
* Clinically significant cardiac disorders (e.g., poorly controlled hypertension, recent MI or stroke, prolonged QTc).
* History or suspicion of interstitial lung disease requiring treatment.
* Active or uncontrolled infection (e.g., hepatitis B with detectable HBV DNA, hepatitis C, HIV, active TB).
* Severe GI conditions impairing drug absorption (e.g., Crohn's, ulcerative colitis).
* Use of strong CYP3A inducers/inhibitors within 1 week or ongoing need for warfarin.
* Participation in another interventional trial within 4 weeks or receipt of a live vaccine within 180 days.
* Any condition that may compromise adherence or safety, per investigator judgment.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 270 (Estimated)
Dates: Start 2025-05 (Estimated); Primary Completion 2030-12 (Estimated); Study Completion 2035-12 (Estimated)

PRIMARY OUTCOMES:
Disease-Free Survival (DFS) | From randomization until disease recurrence or death (up to approximately 5 years)
  Disease-free survival (DFS) is defined as the time from randomization to the first documented disease recurrence (local relapse or distant metastasis confirmed by imaging or pathology) or death from any cause, whichever occurs first. Participants without documented recurrence or death at the time of analysis will be censored at their last disease assessment date.

SECONDARY OUTCOMES:
Overall Survival (OS) | From randomization to death or last follow-up (up to approximately 5 years)
  Overall survival (OS) is defined as the time from randomization to death from any cause. Participants who remain alive or are lost to follow-up at the time of analysis will be censored at the date of last contact.
Central Nervous System Disease-Free Survival (CNS DFS) | From randomization until CNS progression or death, whichever occurs first (up to approximately 5 years)
  CNS DFS is defined as the time from randomization to the date of first occurrence of central nervous system (CNS) metastases or death from any cause, whichever occurs first, as determined by imaging or clinical assessment. Participants without a CNS event or death at the time of analysis will be censored at their last disease assessment date.
Incidence of Treatment-Emergent Adverse Events [Safety and Tolerability] | From date of randomization up to approximately 5 years
  AEs graded by CTCAE version 5.0

IPD SHARING:
Plan to Share IPD: No